CLINICAL TRIAL: NCT01633866
Title: Pediatric Radio Frequency Coil Development on Clinical and Research MR Scanners
Brief Title: Pediatric Radio Frequency Coils Generic
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-1041
Record Dates: First submitted 2012-06-21; First posted 2012-07-04 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Duchenne Muscular Dystrophy; Musculoskeletal Abnormalities
Keywords: Magnetic Resonance Imaging
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Musculoskeletal Abnormalities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Advances in Radio Frequency for MRI: advances in radio frequency (RF) coil magnetic resonance imaging (MRI)

SUMMARY:
The purpose of this study is to evaluate and optimize advances in radio frequency (RF) coil magnetic resonance imaging (MRI) technology at Cincinnati Children's Hospital Medical Center (CCHMC).

DETAILED DESCRIPTION:
Pediatric Magnetic resonance (MR) imaging techniques have been limited by the unavailability of specialized radio-frequency (RF) coils for pediatric imaging. Typically, MR coils are designed for general purpose adult imaging and lack the mechanical design, flexibility and high channel count needed for pediatric imaging. Furthermore, pediatric patients are often positioned decubitus or prone rather than supine. This makes coil positioning even more challenging and often results in images with low SNR and poor image quality. Many coils used in clinical practice have fixed dimensions that do not fit within the realm of "one-size fits all," especially for the huge variation found in the pediatric patient population.

MRI coil development and optimization is performed by MR manufacturers and in research laboratories across the world including the Imaging Research Center (IRC) of Cincinnati Children's Hospital and Medical Center (CCHMC). Coil development and refinement involves evaluating the new coils on inert phantoms and then imaging examinations performed on healthy participants and patients. The focus of this study protocol is to evaluate the design and performance of investigational coils on patients and healthy participants.

ELIGIBILITY:
Inclusion Criteria:

Healthy participants:

* Male or Female
* Thermally stable
* Any age

Clinical patients:

* Male or Female
* Thermally stable
* any age

Exclusion Criteria:

Healthy participants & Clinical patients

* Female participants who are pregnant or lactating
* Subjects iwth standard contraindications to MRI

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy participants will be recruited by word-of-mouth, generally from within CCHMC.The healthy participants could include children of faculty or staff members of CCHMC.Because the healthy participants could include children of faculty or staff members, recruitment will be consistent with CCHMC Research Policy.Patients will be recruited at the time of their scheduled clinical scan.We are only using these participants to evaluate the safety and feasibility of the use of the new coils in our patient population.For this reason, we will not focus on the demographics of the participants.However, we will attempt to obtain a broad anatomic size range to match that of the patient population for which the coils were developed.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2012-07; Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as measured by heating and comfort participant response | Day 1

SECONDARY OUTCOMES:
MRI Image Quality | 2 Weeks Post MRI Scan

CONTACTS AND LOCATIONS:
Overall Officials: Charles Dumoulin, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's, Cincinnati, Ohio, United States